CLINICAL TRIAL: NCT03193086
Title: The Effect of Alemtuzumab on the Blood-brain-barrier and Cerebral Metabolism in Multiple Sclerosis Patients; a New MRI Method for Treatment Response Evaluation in Multiple Sclerosis
Brief Title: The Effect of Alemtuzumab on the Blood-brain-barrier and the Brain's Metabolism in Multiple Sclerosis Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Principal Investigator, Peter FredSvan, Medical Doctor, Glostrup University Hospital, Copenhagen
Other Study IDs: GZ-2016-11629
Record Dates: First submitted 2017-06-14; First posted 2017-06-20 (Actual); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Blood-Brain-Barrier; Treatment response; Metabolism; Alemtuzumab; Perfusion; Oxygen consumption
MeSH Terms: conditions — Multiple Sclerosis | interventions — Alemtuzumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma, urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Alemtuzumab treated MS patients: Those with Multiple Sclerosis that have commenced therapy with alemtuzumab (60 mg infusion over the course of 5 days) and completed treatment with alemtuzumab (additional 36 mg infusion during the course of 3 days, 12 months later).
  Interventions: Drug: Alemtuzumab

INTERVENTIONS:
Drug: Alemtuzumab — Alemtuzumab is administered to eligible patients in accordance with established treatment regimes. Initially 60 mg of alemtuzumab is injected intravenously over the course of 5 days. The first treatment series is followed by the injection of 36 mg of alemtuzumab over the course of 3 days 12 months later. During both drug interventions, the transient exacerbation in disease severity is alleviated by concomitant steroid therapy.
  Other Names: Lemtrada

SUMMARY:
The development and progression of multiple sclerosis seem to be driven by concomitant inflammation and, to a less well-defined degree, disturbances in metabolism of individual cells of the human central nervous system as well as changes in the dynamical supply of blood to the brain. These alterations in normal physiology can be quantified by investigating the change in specific parameters over the time course of multiple sclerosis evolution. Amongst these specific parameters, the ability of the so-called blood-brain-barrier to selectively filter nutrients from the blood stream prior to passage into the nervous tissue, is disrupted in multiple sclerosis, and the severity of this deficiency seem to be related to the underlying disease burden. The present study utilises a novel imaging technology in order to monitor changes in the integrity of the blood-brain-barrier over the course of treatment with a biological disease modifying agent known as alemtuzumab. Alemtuzumab is a potent immunosuppressant drug. It is hypothesised that alemtuzumab reverts the deficiency in blood-brain-barrier integrity and, conversely, the severity of blood-brain-barrier disruption at several time points during alemtuzumab treatment can be utilised as prognostic marker for the requirement of additional administration of alemtuzumab beyond the regular treatment regimen. In addition, several other factors are investigated by advanced imaging techniques in combination with blood and urine samples in order to elucidate the possible underlying mechanism of alemtuzumab efficacy. It is hypothesized that alemtuzumab normalises metabolic alterations and changes in the blood supply through resolution of inflammation in the brains of multiple sclerosis patients.

DETAILED DESCRIPTION:
Traditional paraclinical measures of disease severity in multiple sclerosis (MS), such as T2 lesion load as measured by magnetic resonance imaging (MRI), are poorly correlated with long-term disability accumulation. Other surrogate markers of the current and future disease burden are therefore needed. The permeability of the blood-brain-barrier (BBB) seems to better reflect the substantial, subclinical disease activity underlying MS progression. Its useful role as a prognostic marker in MS has been clearly established by the recent observation that BBB permeability increase in optic neuritis patients is associated with conversion to definite MS. BBB permeability can be quantified, in a convenient manner to the patient, using Dynamic-Contrast-Enhanced Magnetic Resonance Imaging (DCE-MRI) by modelling the change in intrinsic MRI parameters of the human brain in response to the administration of a bolus contrast agent. Alemtuzumab is a disease modifying drug that depletes T- and B-cells. It is administered in two series separated by 12 months, as explained in the section "Groups and Interventions." The number of relapses are significantly reduced as compared to other efficacious treatments in MS, as demonstrated recently (study referred to by its ClinicalTrials.gov identifier NCT00050778). The efficacy of alemtuzumab in resolving the inflammatory burden underlying relapses is, thus, well-established. Its influence on subclinical inflammation, however, remains unknown. It is the aim of the present study to investigate whether or not the latter influence is of importance, and, consequently, can be used to evaluate the need for an intensified treatment, in the form of an additional series of alemtuzumab administration.

BBB permeability changes, as surrogate markers of subclinical inflammation, are measured every 6 months just prior to and during the course of alemtuzumab treatment. In order to elucidate other potential mechanisms involved in disability accumulation, biomarkers and MRI-derived parameters are evaluated concomitantly. Specifically, the role of metabolic changes are investigated using MRI methods that measures blood perfusion and oxygen consumption. Secondarily, the BBB permeability and metabolic changes are correlated to novel biomarkers of inflammation and neurodegeneration in serum and urine, as well as conventional measures of MS severity: annual relapse rate, Expanded Disability Severity Score, MRI-derived estimates of disease activity and brain atrophy.

35 patients are included in the study in order to achieve enough statistical power and accommodate drop-outs. Patients are MRI scanned at baseline, 6 months after alemtuzumab treatment, and, finally, prior to administration of the second series of alemtuzumab 12 months after the baseline MRI scanning. At each time point, the patient's disease status is evaluated by an experienced neurologist, and urine and serum samples are obtained. Repeated Measures Analysis Of Variance (ANOVA) will be used to evaluate changes of permeability of the BBB and metabolic parameters at different time points, and baseline characteristics, such as prednisolone treatment will be implemented as between-subjects covariates. Logistic regression will be applied to estimate the ability of BBB permeability changes to predict the need for additional series of alemtuzumab administration.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of Relapsing-Remitting Multiple Sclerosis
* Eligible for alemtuzumab treatment at Glostrup Hospital or The Danish Kingdom Hospital
* Subjects must be deemed physically and mentally able to participate in the study

Exclusion Criteria:

* Contraindications to MRI scanning (pregnancy, pacemakers, claustrophobia, extreme obesity)
* Contraindications to the use of MRI contrast agents (kidney disease, previous allergic reactions)
* Conflicting disorders (e.g. disorders with a systemic, inflammatory component)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients are recruited from the two dedicated MS clinics in the secondary health care sector of the danish capital region.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-03-31 (Estimated); Study Completion 2020-03-31 (Estimated)

PRIMARY OUTCOMES:
Blood-Brain-Barrier Permeability | 1 year
  Blood-Brain-Barrier Permeability as measured by Dynamic-Contrast-Enhanced MRI (DCE-MRI)

SECONDARY OUTCOMES:
Oxygen Consumption | 1 year
  The Cerebral Metabolic Rate of Oxygen Consumption as measured by a novel MRI technique
Cerebral perfusion | 1 year
  Quantification of cerebral perfusion using DCE-MRI and Arterial-Spin-Labelling MRI
Diffusion Tensor MRI parameters and MR spectroscopy metabolite concentrations | 1 year
  Measurement of changes in microstructural organization as measured by Diffusion Tensor MRI
Brain atrophy | 2 years
  Voxel-Based-Morphometry of grey and white matter utilizing high-resolution MRI
Clinical Severity of Disease | 1 year
  Estimation of disease severity by the Expanded Disability Severity Scale (EDSS)
Relapse frequency | 1 year
  Number of relapses during follow-up and past history
Plasma markers of Blood-Brain-Barrier breakdown | 1 year
  Detection of markers associated with Blood-Brain-Barrier breakdown nervous system
Plasma markers of neuronal damage | 1 year
  Detection of markers associated with neuronal damage
Urinary markers of inflammation | 1 year
  Detection of markers associated with inflammatory activity specific to macrophages/microglia in the human central nervous system

CONTACTS AND LOCATIONS:
Overall Officials: Henrik BW Larsson, MD, Prof., Study Director — Functional Imaging Unit, Department of Clinical Physiology, Nuclear medicine and PET, Glostrup Hospital
Locations (1):
- Functional Imaging Unit, Department of Clinical Physiology, Nuclear medicine and PET, Glostrup Hospital, Glostrup Municipality, Copenhagen Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barkhof F. The clinico-radiological paradox in multiple sclerosis revisited. Curr Opin Neurol. 2002 Jun;15(3):239-45. doi: 10.1097/00019052-200206000-00003. PMID 12045719
- [Background] Cramer SP, Larsson HB. Accurate determination of blood-brain barrier permeability using dynamic contrast-enhanced T1-weighted MRI: a simulation and in vivo study on healthy subjects and multiple sclerosis patients. J Cereb Blood Flow Metab. 2014 Oct;34(10):1655-65. doi: 10.1038/jcbfm.2014.126. Epub 2014 Jul 30. PMID 25074746
- [Background] Broholm H, Andersen B, Wanscher B, Frederiksen JL, Rubin I, Pakkenberg B, Larsson HB, Lauritzen M. Nitric oxide synthase expression and enzymatic activity in multiple sclerosis. Acta Neurol Scand. 2004 Apr;109(4):261-9. doi: 10.1111/j.1600-0404.2004.00207.x. PMID 15016008
- [Background] Cramer SP, Modvig S, Simonsen HJ, Frederiksen JL, Larsson HB. Permeability of the blood-brain barrier predicts conversion from optic neuritis to multiple sclerosis. Brain. 2015 Sep;138(Pt 9):2571-83. doi: 10.1093/brain/awv203. Epub 2015 Jul 17. PMID 26187333
- [Background] D'haeseleer M, Cambron M, Vanopdenbosch L, De Keyser J. Vascular aspects of multiple sclerosis. Lancet Neurol. 2011 Jul;10(7):657-66. doi: 10.1016/S1474-4422(11)70105-3. PMID 21683931
- [Background] Gauthier SA, Berger AM, Liptak Z, Duan Y, Egorova S, Buckle GJ, Glanz BI, Khoury SJ, Bakshi R, Weiner HL, Guttmann CR. Rate of brain atrophy in benign vs early multiple sclerosis. Arch Neurol. 2009 Feb;66(2):234-7. doi: 10.1001/archneurol.2008.567. PMID 19204160
- [Background] Ge Y, Zhang Z, Lu H, Tang L, Jaggi H, Herbert J, Babb JS, Rusinek H, Grossman RI. Characterizing brain oxygen metabolism in patients with multiple sclerosis with T2-relaxation-under-spin-tagging MRI. J Cereb Blood Flow Metab. 2012 Mar;32(3):403-12. doi: 10.1038/jcbfm.2011.191. Epub 2012 Jan 18. PMID 22252237
- [Background] De Keyser J, Steen C, Mostert JP, Koch MW. Hypoperfusion of the cerebral white matter in multiple sclerosis: possible mechanisms and pathophysiological significance. J Cereb Blood Flow Metab. 2008 Oct;28(10):1645-51. doi: 10.1038/jcbfm.2008.72. Epub 2008 Jul 2. PMID 18594554
- [Background] Larsson HB, Stubgaard M, Frederiksen JL, Jensen M, Henriksen O, Paulson OB. Quantitation of blood-brain barrier defect by magnetic resonance imaging and gadolinium-DTPA in patients with multiple sclerosis and brain tumors. Magn Reson Med. 1990 Oct;16(1):117-31. doi: 10.1002/mrm.1910160111. PMID 2255233
- [Background] Larsson HB, Courivaud F, Rostrup E, Hansen AE. Measurement of brain perfusion, blood volume, and blood-brain barrier permeability, using dynamic contrast-enhanced T(1)-weighted MRI at 3 tesla. Magn Reson Med. 2009 Nov;62(5):1270-81. doi: 10.1002/mrm.22136. PMID 19780145
- [Background] Law M, Saindane AM, Ge Y, Babb JS, Johnson G, Mannon LJ, Herbert J, Grossman RI. Microvascular abnormality in relapsing-remitting multiple sclerosis: perfusion MR imaging findings in normal-appearing white matter. Radiology. 2004 Jun;231(3):645-52. doi: 10.1148/radiol.2313030996. PMID 15163806
- [Background] Naismith RT, Cross AH. Enhancing our understanding of white matter changes in early multiple sclerosis. Brain. 2015 Sep;138(Pt 9):2465-6. doi: 10.1093/brain/awv196. No abstract available. PMID 26304148
- [Background] Scalfari A, Neuhaus A, Degenhardt A, Rice GP, Muraro PA, Daumer M, Ebers GC. The natural history of multiple sclerosis: a geographically based study 10: relapses and long-term disability. Brain. 2010 Jul;133(Pt 7):1914-29. doi: 10.1093/brain/awq118. Epub 2010 Jun 9. PMID 20534650
- [Background] Steen C, D'haeseleer M, Hoogduin JM, Fierens Y, Cambron M, Mostert JP, Heersema DJ, Koch MW, De Keyser J. Cerebral white matter blood flow and energy metabolism in multiple sclerosis. Mult Scler. 2013 Sep;19(10):1282-9. doi: 10.1177/1352458513477228. Epub 2013 Feb 21. PMID 23428956
- [Background] Sun X, Tanaka M, Kondo S, Okamoto K, Hirai S. Clinical significance of reduced cerebral metabolism in multiple sclerosis: a combined PET and MRI study. Ann Nucl Med. 1998 Apr;12(2):89-94. doi: 10.1007/BF03164835. PMID 9637279
- [Background] Tuohy O, Costelloe L, Hill-Cawthorne G, Bjornson I, Harding K, Robertson N, May K, Button T, Azzopardi L, Kousin-Ezewu O, Fahey MT, Jones J, Compston DA, Coles A. Alemtuzumab treatment of multiple sclerosis: long-term safety and efficacy. J Neurol Neurosurg Psychiatry. 2015 Feb;86(2):208-15. doi: 10.1136/jnnp-2014-307721. Epub 2014 May 21. PMID 24849515
- [Background] Coles AJ, Fox E, Vladic A, Gazda SK, Brinar V, Selmaj KW, Skoromets A, Stolyarov I, Bass A, Sullivan H, Margolin DH, Lake SL, Moran S, Palmer J, Smith MS, Compston DA. Alemtuzumab more effective than interferon beta-1a at 5-year follow-up of CAMMS223 clinical trial. Neurology. 2012 Apr 3;78(14):1069-78. doi: 10.1212/WNL.0b013e31824e8ee7. Epub 2012 Mar 21. PMID 22442431